CLINICAL TRIAL: NCT06667726
Title: A Centralized Protocol Evaluating the Safety and Clinical Impact of Amino Acid Pet for Brain Tumors
Brief Title: An Investigational Scan (18F-DOPA PET/CT) for Improving the Clinical Management of Brain Tumors
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 24-000426; NCI-2024-08915 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-000426 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Malignant Brain Neoplasm
MeSH Terms: conditions — Brain Neoplasms | interventions — fluorodopa F 18; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (18F-DOPA) (Experimental): Patients receive 18F-DOPA IV and undergo PET/CT over 30 minutes on day 1.
  Interventions: Procedure: Computed Tomography; Drug: Fluorodopa F 18; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Fluorodopa F 18 — Given IV
  Other Names: (18F)FDOPA; 18F-DOPA; 18F-FDOPA; 3-(2-Fluoro-(sup 18)F-4,5-dihydroxyphenyl)-L-alanine; 6-(18F)Fluoro-L-DOPA; Fluorine F 18 Fluorodopa; Fluorine-18-fluoro-L-DOPA; Fluorodopa (18F); FLUORODOPA F-18; L-6-(18F)Fluoro-DOPA
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT

SUMMARY:
This phase II trial studies how well the addition of 18F-DOPA (amino acid) positron emission tomography (PET)/computed tomography (CT) to standard of care (SOC) imaging can improve the clinical management of patients with brain tumors in over 50% of cases. PET is an imaging test that helps to measure the information about functions of tissues and organs within the body. A PET scan uses a radioactive drug (radiotracer) to show this activity. CT scan uses X-rays to create images of the bones and internal organs within the body. Combining a PET scan with a CT scan can help make the images easier to interpret. PET/CT scans are hybrid scanners that combine both of the two modalities into a single scan. This allows images of both anatomy (CT) and function (PET) to be taken during the same scan. The 18F-DOPA PET/CT scan is done with a very small amount of a radioactive tracer called FDOPA. The PET/CT scan is then used to detect the location of tumors. Using the 18FDOPA-PET/CT scan in addition to the SOC scan may improve the clinical management of patients with brain tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether the addition of amino acid PET to standard of care imaging impacts clinical management of brain tumor patients in over 50% of cases.

SECONDARY OBJECTIVES:

I. To assess the safety and tolerability of amino acid PET for brain tumor patients in response to Food and Drug Administration (FDA) guidance that such data is needed to support a potential New Drug Application (NDA) for fluorodopa F 18 (18F-DOPA).

II. To assess the rate of identification of tumor outside of standard magnetic resonance imaging (MRI) imaging.

OUTLINE:

Patients receive 18F-DOPA intravenously (IV) and undergo PET/CT over 30 minutes on day 1.

After completion of study intervention, patients are followed for 3 days.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Diagnosis of a brain tumor
* Indication for amino acid PET imaging, including presurgical evaluation, radiation planning, MR imaging indeterminate for progression versus treatment effect, or clinical need for enhanced monitoring
* Ability to give appropriate consent or have an appropriate representative available to do so

Exclusion Criteria:

* Patient is unable to undergo PET imaging
* Persons who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2029-10-08 (Estimated); Study Completion 2029-10-08 (Estimated)

PRIMARY OUTCOMES:
Impact of 18F-DOPA PET/CT on clinical management | 3 days post-PET scan, up to 64 days
  Will be measured using the Amino Acid PET Imaging Survey, to be completed by the provider after participant has received fluorodopa F 18 (18F-DOPA) positron emission tomography (PET)/computed tomography (CT). The survey consists of 4 questions, 1 multiple choice (what will PET scan be used for); 2 yes/no and one open-ended question related with how PET scan did or did not make a clinically meaningful impact in the management of patient care.

SECONDARY OUTCOMES:
Incidence of adverse events | 3 days post-PET scan, up to 64 days
  Will be assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Rate of identification of tumor outside of standard magnetic resonance imaging (MRI) | 3 days post-PET scan, up to 64 days
  Will be measured using the Amino Acid PET Imaging Survey, to be completed by the provider after participant has received fluorodopa F 18 (18F-DOPA) positron emission tomography (PET)/computed tomography (CT). The survey consists of 4 questions, 1 multiple choice (what will PET scan be used for); 2 yes/no (including whether a tumor outside of MRI contrast enhancement was identified); and one open-ended question related with how PET scan did or did not make a clinically meaningful impact in the management of patient care.

CONTACTS AND LOCATIONS:
Overall Officials: Derek R. Johnson, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials